CLINICAL TRIAL: NCT02080702
Title: An International, Multicentric, Prospective, Observational Study to Evaluate Monosyn® Suture Material for Anastomoses in the Gastrointestinal Tract.
Acronym: PROMEGAT
Status: Terminated | Type: Observational
Why Stopped: Planned recruitment of 630 patients was not possible to achieve within the given time frame
Sponsor: Aesculap AG (Industry)
Collaborators: B.Braun Surgical SA (Industry)
Responsible Party: Sponsor
Other Study IDs: AAG-O-H-1209
Record Dates: First submitted 2014-03-05; First posted 2014-03-06 (Estimated); Last update posted 2018-07-02 (Actual); Status verified 2018-06

CONDITIONS: C.Surgical Procedure; Digestive System; Symptomatic Disorders of the Gastrointestinal Tract; Gastric Anastomosis (Site); Gastrointestinal Neoplasms
Keywords: GIT, Monosyn, anastomoses leakage
MeSH Terms: conditions — Gastrointestinal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Monosyn: Construction of a gastrointestinal anastomoses
  Interventions: Device: Monosyn

INTERVENTIONS:
Device: Monosyn — Monosyn will be used to perform the gastrointestinal anastomoses

SUMMARY:
The aim of this non-interventional study is to evaluate the efficacy of a monofilament, mid-term absorbable suture material (Monosyn®) for anastomosis performed in the gastrointestinal tract using the frequency of anastomosis leakage as a primary parameter.

Postoperative complication rate, length of hospital stay, costs, time to perform the anastomosis and handling will serve as secondary endpoints.

The question is addressed, whether a monofilament suture material is as effective as a braided suture material for anastomosis construction within the gastrointestinal tract.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years and older
* ASA I-III
* Indication for an elective tumor surgery within the GI tract (stomach, small intestine, large intestine)
* Written informed consent

Exclusion Criteria:

* Emergency surgery
* Peritonitis
* Patients undergoing an operation due to a tumour within the pancreas, rectum, esophagus
* Pregnant women and breast-feeding women
* Chemotherapy
* Current immunosuppressive therapy
* Radiotherapy on the treated region within the last 2 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult patients
Sampling Method: Non-Probability Sample
Enrollment: 106 (Actual)
Dates: Start 2014-08; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Frequency of anastomosis leakage rate | participants will be followed for the duration of hospital stay, an expected average of 7 days
  Anastomotic leak is defined as radiographic demonstration of a fistula or non-absorbable material drainage from a wound after oral administration, or visible disruption of the suture line during re-exploration.

SECONDARY OUTCOMES:
Postoperative complication rate | participants will be followed for the duration of hospital stay, an expected average of 7 days
  As postoperative complications the following parameter will be documented: peritonitis, wound infection, bleeding, abscess, fistula, perforation, obstipation and stenosis. Wound infections, peritonitis and abscess are defined according to the Centres for Disease Control and Prevention (CDC, 17).
Reoperation rate | participants will be followed for the duration of hospital stay, an expected average of 7 days
Length of hospital stay | participants will be followed for the duration of hospital stay, an expected average of 10 days
  Duration from day of operation until the day of discharge from the hospital.
Stay in the intensive care unit | participants will be followed for the duration of hospital stay, an expected average of 7 days
  Duration from the first day in the ICU until the last day in the ICU. In the case of readmission to the ICU the sum of all days within the ICU.
Duration to perform the anastomosis | intraoperatively
  The time recorded for the construction of the anastomosis begins with the placement of the first stitch and ends with cutting the excess material from the last stitch.
Cost | duration of the intervention (approximately 18 months)
  Calculation of the cost of material is based on the actual hospital costs for the suture material and the number of used threads by the surgeon.
  For the calculation of the operation costs, the time to perform the anastomosis will be multiplied with the cost of one operation minute (50-100 €).
Handling of the device | End of the Study (approximately 18 months)
  Intra-operative handling of the suture material will be reported on a separate document one time per participating surgeon at the end of the study. The following criteria will be assessed:
  knot security, knot pull tensile strength, knot run-down, tissue drag, elasticity and feeling of the suture material. For the rating a 5-point scale is used

CONTACTS AND LOCATIONS:
Locations (5):
- University Malaya Medical Centre, Kuala Lumpur, Malaysia
- Philippine General Hospital, Manila, Philippines
- South Korea (2):
  - GangNam Severance Hospital, Gangnam-Gu, Seoul
  - Seoul National University Bundang Hospital, Gyeonggi-do
- Veterans General Hospital-Taipei, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Baumann P, Kim J, Ahn SH, Kim HH, Chong HY, Wente MN. Mid-term absorbable monofilament is safe and effective for gastrointestinal anastomosis - PROMEGAT - A single-arm prospective observational study. Ann Med Surg (Lond). 2018 Apr 6;30:1-6. doi: 10.1016/j.amsu.2018.04.003. eCollection 2018 Jun. PMID 29946452